CLINICAL TRIAL: NCT01243723
Title: Étude Comparative, randomisée, Double-insu, en Groupes parallèles évaluant l'efficacité d'Eductyl® Versus Placebo Chez Des Patients Souffrant d'Une dyschésie
Brief Title: Study Assessing the Efficacy of Eductyl® for the Treatment of Patients With Dyschesia
Acronym: EDUCDYS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratoires Techni Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010-021919-17
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Dyschesia
Keywords: Dyschesia treatment; Inconfort related to dyschesia; Quality of life; Bowel function index
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eductyl suppository (Experimental)
  Interventions: Drug: Eductyl suppository
- Placebo suppository (Placebo Comparator)
  Interventions: Drug: Placebo suppository

INTERVENTIONS:
Drug: Eductyl suppository — One suppository every morning during 21 days
  Arms: Eductyl suppository
Drug: Placebo suppository — One suppository every morning during 21 days
  Arms: Placebo suppository

SUMMARY:
The purpose of this study is to assess the efficacy of Eductyl versus placebo for treatment of patients with dyschesia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged from 18 to 75 years old,
* Writing consent to take part in the study,
* Patient with a dyschesia according to Rome III criteria
* An intensity of the inconfort using a VAS (0 (no inconfort) to 100 mm (maximal and no supportable inconfort)) equal or over 40 mm

Exclusion Criteria:

* Patient suffering of neurologic affection,
* Rectal diseases including :

  * Current anal ou peri-anal pain,
  * Current organic injury of colon or rectum,
  * Current anal injury,
  * Current rectal Prolapse,
  * Current haemorrhoid,
  * Colon inflammatory disease (ulcero haemorrhagic recto colitis, Crohn disease…),
  * Current ano-recto-colon stenosis (anastomosis, scarring ...)
* Patient undergone pain killers (WHO level II (except dextropropoxyphen) and III) during the last 8 days,
* Patient undergone anti-depressants except if this treatment is regular for at least 15 days and it won't be modified during the study,
* Patient with a constipation treatment except if this treatment is regular for at least 15 days and it won't be modified during the study
* Intolerance to Eductyl® or to one of its components (potassium tartarate acid, sodium bicarbonate, solid hemisynthethic glycerides, soya lecithin, talc)
* Use of Eductyl® during the previous 15 days (over 5 days in the last 15 days),
* Patient already included in clinical trial in the last month,
* Pregnant or breast feeding woman,
* Woman of childbearing potential without contraception,
* Patient unable to read and write.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2010-11; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of Eductyl versus placebo for treatment of patients with dyschesia on VAS of intensity of inconfort | Day 0 and day 21

SECONDARY OUTCOMES:
To assess the intensity of inconfort of patients with dyschesia on Likert scale | Every day from day 0 to day 21
To assess the efficacy of Eductyl versus placebo on dyschesia related quality of life | Day 0 and day 21
To assess the efficacy of Eductyl versus placebo on bowel function index | Day 0 and day 21
To assess the efficacy of Eductyl versus placebo on global impression of change | Day 21
To assess the tolerance of Eductyl versus placebo | Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Laure Tarrerias, Dr, Principal Investigator — Suresnes Hospital; Bernard Savarieau, Dr, Study Director — Nukleus
Locations (1):
- Hôpital Foch, Service de Chirurgie Générale et Digestive, Suresnes, France